CLINICAL TRIAL: NCT04141969
Title: A Novel Nutraceutical to Combat Post-Lyme Disease Syndrome
Acronym: PLDS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Optimal Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RLP10242019
Record Dates: First submitted 2019-10-25; First posted 2019-10-28 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-01

CONDITIONS: Post-Lyme Disease Syndrome (PLDS)
Keywords: Lyme
MeSH Terms: conditions — Post-Lyme Disease Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RLP (Active Comparator): ReaLife+
  Interventions: Dietary Supplement: RLP
- Inert (Placebo Comparator): Inert brown powder to look similar to RLP
  Interventions: Other: Placebo
- Control (No Intervention): Not given RLP or the placebo

INTERVENTIONS:
Dietary Supplement: RLP — RLP nutraceutical
  Arms: RLP
Other: Placebo — Inert brown powder
  Arms: Inert

SUMMARY:
This study will determine the effectiveness of a nutraceutical in treating the lingering effects of Lyme Disease after antibiotic treatment.

DETAILED DESCRIPTION:
A Novel Nutraceutical to Combat Post-Lyme Disease Syndrome will be evaluated during a double blind, placebo controlled study. This study is an expansion of RLP042019 NCT04078841 Treating Post-Lyme Disease Syndrome With Acetogenins

ELIGIBILITY:
Inclusion Criteria:

1. A positive two-test methodology using a sensitive enzyme immunoassay (EIA) or immunofluorescence assay as a first test, followed by a western immunoblot assay for specimens yielding positive or equivocal results for Lyme Disease that has been treated with antibiotics but the symptoms persist post treatment.
2. Must be able to swallow a mixed powder drink.

Exclusion Criteria:

1 .Non Positive Western Blot test.

2. Positive Western Blot test where the individual has not been treated with antibiotics.

-

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-28 (Actual)

PRIMARY OUTCOMES:
PROMIS Global-10 | 6 months
  PROMIS Global-10; Self reported level changes as measured by the Patient-Reported Outcomes Measurement Information System Global-10 .
IHT Blood Test Assessment | 6 months
  Outcome measure of "positive" or "negative" for antibodies; IgG P93 Ab. IgG P66 Ab. IgG P58 Ab. IgG P45 Ab. IgG P41 Ab. IgG P39 Ab. IgG P30 Ab. IgG P28 Ab. IgG P23 Ab. IgG P18 Ab.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Osguthorpe, ND, Principal Investigator — Optimal Health Research
Locations (1):
- Optimal Health Research, Salt Lake City, Utah, United States